CLINICAL TRIAL: NCT03929848
Title: Minimum Cuff Pressure to Prevent Gas Leakage During Mechanical Ventilation in Laryngomicrosurgery - Pilot Study -
Brief Title: Cuff Pressure in LMS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-2018-106
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Laryngomicrosurgery
Keywords: cuff pressure, laryngomicrosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- female: female patient who is scheduled for laryngomicrosurgery
  Interventions: Procedure: Cuff pressure
- male: male patient who is scheduled for laryngomicrosurgery
  Interventions: Procedure: Cuff pressure

INTERVENTIONS:
Procedure: Cuff pressure — observe and record the required cuff pressure to prevent gas leakage during mechanical ventilation for laryngomicrosurgery

SUMMARY:
The goal of this prospective observational study is to investigate minimum cuff pressure to prevent gas leakage during mechanical ventilation in laryngomicrosurgery.

DETAILED DESCRIPTION:
It has been well known that cuff pressure should be adequately limited to prevent ischemic injury of tracheal mucosa, which is about 20-30 mmHg. However, higher cuff pressure that 20-30 mmHg might be required to prevent gas leakage during general anesthesia for laryngomicrosurgery.

The hypothesis of this study is that the required cuff pressure to prevent gas leakage from mechanical ventilation during general anesthesia for laryngomicrosurgery, and there will be no damage from the required cuff pressure because of short time of surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients who is scheduled for laryngomicrosurgery due to simple vocal cord cyst or nodule

Exclusion Criteria:

* Who doesn't agree to enroll
* do not use a reinforced tracheal tube of internal diameter of 5.5 mm for male patient
* do not use a reinforced tracheal tube of internal diameter of 5.0 mm for female patient

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient who is scheduled for laryngomicrosurgery due to simple vocal cord cyst or nodule
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2019-04-30 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Cuff pressure | intraoperative
  the required cuff pressure to prevent gas leakage from mechanical ventilation during general anesthesia for laryngomicrosurgery
post operative complication | from end of surgery to 1-2 weeks after surgery
  any postoperative symptoms associated with cuff pressure such as hoarsness, dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Man Lee, M.D.,PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea